CLINICAL TRIAL: NCT05486676
Title: VR-Moodboost in the Treatment of Depression; a Proof-of-concept Study
Brief Title: VR-Moodboost; an Innovative Virtual Reality Treatment for Adolescents With Depression
Acronym: VR-Moodboost
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Claudi Bockting (Other)
Collaborators: GGZ Delfland (Unknown)
Responsible Party: Sponsor-Investigator, Claudi Bockting, Professor of Clinical Psychology in Psychiatry, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77018.018.21
Record Dates: First submitted 2022-07-25; First posted 2022-08-03 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Virtual Reality; Positive affect; Depressive symptoms; Adolescents
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: The study has a non-concurrent, multiple baseline, single-case, AB-design. Participants will first be randomly allocated to a 3 or 5-week baseline period. After baseline (A-phase), a trained therapist performs the 12 session VR-Moodboost (B-phase).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-Moodboost (Experimental): All participants receive the same VR-Moodboost treatment, they only differ in the length of the baseline; 3 or 5 weeks.
  Interventions: Behavioral: VR-Moodboost; a Virtual Reality intervention for depression to enhance positive affect and reduce depressive symptoms.

INTERVENTIONS:
Behavioral: VR-Moodboost; a Virtual Reality intervention for depression to enhance positive affect and reduce depressive symptoms. — All participants receive the same VR-Moodboost treatment, they only differ in the length of the baseline; 3 or 5 weeks.

SUMMARY:
Major depressive disorder (MDD) is a prevalent and disabling mental health condition. A recent meta-analysis shows that across all forms of psychotherapy, only 43% of all depressive patients fully recover from MDD and relapse rates are high. Therefore, there is a strong need for innovative interventions with better treatment outcomes. Most traditional psychotherapies for depression focus on reducing negative affect. However, in patients suffering from depression, anhedonia, or loss of positive affect, is associated with poor prognosis and increased chance of suicide. Recent studies show promising results for novel psychotherapies with a focus on enhancing positive affect. Experimental studies indicate that non-verbal stimuli have a stronger impact on activation of positive affect than verbal stimuli, which makes Virtual reality (VR) a promising tool to enhance positive affect. For the current study the investigators developed an innovative VR treatment protocol to enhance positive affect and reduce depressive symptoms in patients with MDD.

This study will include 10 adolescents aged 15 to 23 years old, who have a diagnosis of unipolar mild to severe depression. A trained psychologist will perform the VR-Moodboost intervention in twelve weekly sessions.

The overall aim of this explorative proof-of-concept study is to provide first evidence that treatment with VR-Moodboost will lead to symptom improvement in adolescents with depression. The investigators hypothesize that VR-Moodboost will lead to an increase in positive affect, daily positive mood and a decrease in negative affect and daily negative mood in adolescents with mild to severe depression. Secondary, the investigators hypothesize that the VR-moodboost will lead to a decrease of depressive symptoms, an increase in daily activation, an increase in quality of life and an increase of self-efficacy for the participating patients. Moreover, the investigators hypothesize that VR-Moodboost leads to high patient acceptability and high usability for both patient and therapist.

DETAILED DESCRIPTION:
Adolescents with a depressive disorder who might be eligible for participation will be asked for permission to be contacted by a researcher by their treating psychologist or treating physician either face-to-face, by telephone or by e-mail. Researchers will inform the potential participants about the study by means of a patient information letter and the possibility to ask additional questions by telephone or in a face to face appointment with the researcher. The participant must sign informed consent before participation. The potential participant will be given one week to consider their decision to participate in the study.

The population consists of 10 participants. As indicated by the framework 'effectladder' which is used by the Netherlands Youth Institute to determine which interventions are evidence-based, a sample size of N=10 is sufficient to demonstrate evidence if the effect of treatment is replicated in the majority of cases. By using daily diary data in the baseline and treatment phase of the study, we will be able to compare change in symptoms in baseline phase with change in symptoms in treatment phase.

The VR-Moodboost treatment consists of 12 sessions, and in these sessions the Virtual Reality software Social Worlds VR-CBT will be used. Social Worlds VR-CBT has a medical certificate, and has many different treatment possibilities. In this study, the investigators make use of a specific part of the software; a Virtual Reality environment in which participants can perform activities of choice and get rewarded for the activities they did at home. The first session of the VR-Moodboost treatment will start with psychoeducation about depression and about the rationale of the treatment and the main aim; to increase positive affect. Every next session, the patient will perform different virtual activities of choice, for more information about the activities see 'VR environment'. Because the main aim of the VR-Moodboost treatment is to increase positive affect, patients will be supported and encouraged to (learn to) experience positive affect. For example, the patients will be encouraged to label his/her emotions during the activity in VR, and during the discussion of the homework. In addition, cognitive challenge techniques will be used to stimulate patients to pay attention to positive aspects of a situation (for example, mention 3 positive things or aspects in the VR environment). At the end of each session, the therapist encourages the participant to convert the virtual activity practiced during session into a real-life activity, which would evoke the same positive feeling as the virtual activity and will be practiced at home. The patient will be stimulated to visualize this activity as a goal for the upcoming week. Then the next session, after reflecting on the activity the patient did at home, the participant gets a reward in de VR environment. In general, every session has the following structure; reflect on the activity which the patient did in real life, reveal a virtual reward, perform different virtual activities of choice, explore and visualize an activity for the following week. The sixth session includes an evaluation, and the last session includes a relapse prevention plan.

The study has a non-concurrent, multiple baseline, single-case, AB-design. Participants will first be randomly allocated to a 3 or 5-week baseline period as recommended by What Works Clearinghouse (WWC). During the baseline period the patient will make a personal alert plan with their treating psychologist. After baseline (A-phase), a trained therapist performs the 12 session VR-Moodboost (B-phase). The investigators will measure the primary and secondary outcomes at start baseline, start intervention, post intervention and after a 1-month follow-up period. The acceptability of the session will be measured after every session of therapy. During the A- and B-phase, patients will keep track of their daily mood, activities and self-efficacy using a patient diary by means of a smartphone app. After all 10 participants have conducted the B-phase, a focus group will be organized for both the patients and therapists who have participated to obtain feedback about the VR-Moodboost intervention.

The main study parameters are positive and negative affect and daily positive and negative mood. In this proof-of-concept study results will be analyzed at the individual case level in two ways: using questionnaires at 4 time points and using daily diary data. The investigators will calculate the Reliable Change Index to assess statistical significance of differences in questionnaire scores between time points. The Reliable Change Index is calculated as follows: (posttest- pretest)/ SEM, where SEM = SDinstrument * √(1- reliability). Daily diary data will be analyzed using multilevel analysis using Shiny app MultiSCED. At the individual level the investigators assess whether the intercept and slope on positive and negative mood in the baseline phase significantly differs from the intercept and slope in the treatment phase. Results will be aggregated across participants using the meta-analysis method. State of the art of imputation of missings will be used.

The handling of the personal data is according to the Dutch Act on Implementation of the General Data Protection Regulation (in Dutch: Uitvoeringswet AVG, UAVG). The investigators will separate he data files from the name and date of birth files. The name and date of birth file will be locked with a password; this file contains a code for each participant. The code is a three-digit patient number (YYY). The data files will be collected in the online database Castor. The coordinating investigators safeguard the key to the code. Data will be kept for 15 years according to the aforementioned act.

The Amsterdam UMC Clinical Monitoring Center (CMC) will monitor this study according to the guidelines of the Dutch Federation of University Medical Centres (NFU: Nederlandse Federatie van Universitaire Medische Centra). The CMC-CRA prepared a monitoring plan based on the study protocol in agreement with the coordinating investigator.

All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded. The investigator will report all SAEs to the sponsor without undue delay after obtaining knowledge of the events. The sponsor will report the SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 7 days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of 8 days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after the sponsor has first knowledge of the serious adverse events.

ELIGIBILITY:
Inclusion criteria

* A principal diagnosis of mild-severe depression, either a first or a recurrent episode, as determined by a BIG-registered psychologist (clinical or GZ) or psychiatrist. The severity of the current depressive episode will be determined following the guidelines of the SCID-5 and the SCID-5 Junior.
* Age between 15-23.
* Written informed consent by the patient (age 16-23) or by the patients AND a caregiver (age 15) to participate in the study.

Exclusion criteria

* Intellectual disability in the history.
* A principal diagnosis of depression with psychotic features.
* Current high suicidality risk (suicidality plans).
* Severe comorbid psychiatric disorders including schizophrenia-like disorders, bipolar disorder or addictive disorders in the past six months.
* Current use of antidepressants, antipsychotics or sedatives.
* Uncorrected hearing- or vision problems

Ages: 15 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-07-25 (Estimated); Study Completion 2024-07-25 (Estimated)

PRIMARY OUTCOMES:
Change in positive and negative affect, as measured by the Positive and Negative Affect Schedule (PANAS). | There are two different baseline periods; 3 or 5 weeks. This metric is assessed at week 0 (start baseline), at week 3 or 5 (start VR-Moodboost therapy), at week 15 or 17 (study completion), and at week 19 or 21 (follow-up).
  Scores can range from 10-50 for both Positive affect and Negative affect with the lower scores representing lower levels of Positive/Negative Affect and higher scores representing higher levels of Positive/Negative Affect.
Change in Positive and Negative Affect (Smartphone Diary) | Daily, from baseline till end of intervention phase (15-17 weeks)
  Daily positive and negative affected as measured by 3 items for negative and 3 items for positive mood. Items were based on previous daily diary studies. This metric is assessed through a smartphone diary, from start baseline until the end of the VR-Moodboost therapy (15-17 weeks).

SECONDARY OUTCOMES:
BDI-II - Beck Depression Inventory | This metric is assessed at week 0 (start baseline), at week 3 or 5 (start VR-Moodboost therapy), at week 15 or 17 (study completion), and at week 19 or 21 (follow-up).
  Depressive symptoms as measured by the Beck Depression Inventory (BDI-II). The score range is 0 to 63. Higher scores mean more severe depression symptoms.
Activation (Smartphone Diary) | Daily, from baseline till end of intervention phase (15-17 weeks)
  Activation (daily estimation of number of minutes active) as measured with the daily smartphone diary. This metric is assessed through a smartphone diary, from start baseline until the end of the intervention phase (15-17 weeks).
Self-efficacy (Smartphone Diary) | Daily, from baseline till end of intervention phase (15-17 weeks)
  Single item about self-efficacy "Right now, I believe I can succeed my current goals, if I set my mind to it", scored on a 7-point Likert scale.
KIDSSCREEN / WHOQOL-BREF - Quality of life | This metric is assessed at week 0 (start baseline), at week 3 or 5 (start VR-Moodboost therapy), at week 15 or 17 (study completion), and at week 19 or 21 (follow-up).
  Quality of life as measured by the KIDSSCREEN (age 15-17) and the WHOQOL-BREF (age 18-23). Both at the WHOQOL-BREF and the KIDSSCREEN, higher scores mean better quality of life. Score range of the KIDSSCREEN is 27-135. For the WHOQOL-BREF, There is no overall score, each domain is calculated by summation of their specific items. Maximum scores are: Overall quality of life and General health; 20; Physical health; 35, Psychological health 30, Social relationships 15, and Environment; 40.
The General Self-Efficacy Scale (GSES) | This metric is assessed at week 0 (start baseline), at week 3 or 5 (start VR-Moodboost therapy), at week 15 or 17 (study completion), and at week 19 or 21 (follow-up).
  A general sense of perceived self-efficacy as measured with the General Self-Efficacy Scale (GSES).De score range is 10 to 40. Higher scores mean better self-efficacy.
SRS - Session Rating Scale | From week 3 or 5 to week 15 or 17 (weekly at every VR-session)
  Acceptability as measured by the Session Rating Scale (SRS). The score range is 0-40. Higher scores mean better acceptability.
IPQ - I-Group Presence Questionnaire | At week 15 or 17
  Presence in VR as measured by the I-group presence questionnaire (IPQ). Score range is 0-6. A higher score indicating a greater experienced presence in VR.
SUS - System Usability Scale | At week 3 or 5 and week 15 or 17
  Usability as measured by the System Usability Scale (SUS). SUS scores range from 0 to 100, higher scores mean better SUS.
Line of sight in VR | From week 3 or 5 to week 15 or 17 (weekly at every VR-session)
  Line of sight of participants in VR (extent to which the line of sight deviates from a fixed anchor point) to assess active involvement. This metric is assessed during the 12 VR-Moodboost sessions.
Semi-structured Interview | At week 15 or 17 (end of VR-Moodboost therapy)
  Semi-structured interview for both patient and therapist about their experience with the VR-Moodboost. This metric is assessed at the end of the intervention phase.
Focus Group | At the end of study, estimated 1 year.
  Feedback from focus group with participating patients and therapists about their experience, acceptability and usability of the VR-moodboost. This metric is assessed at the end of the intervention phase.

OTHER OUTCOMES:
Demographics & Other | During screening
  Other measures include demographic information, gender, age, level of education, use of medication in addition to diagnosis (mild, moderate, severe, first episode or recurrent). The measures are assessed during the screening.

CONTACTS AND LOCATIONS:
Overall Officials: Claudi LH Bockting, PhD, Principal Investigator — Department of Psychiatry, University of Amsterdam, Amsterdam University Medical Centers, Amsterdam, The Netherlands; Centre for Urban Mental Health, University of Amsterdam, The Netherlands
Locations (1):
- GGZ Delfland, Delft, South Holland, Netherlands